CLINICAL TRIAL: NCT04115410
Title: PD-1 Immune Checkpoint Inhibitors and Immune-Related Adverse Events: a Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sungkyunkwan University (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Ju-Young Shin, Assistant Professor, Sungkyunkwan University
Other Study IDs: SKKU-2019-PD1ICI
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Immune-Related Adverse Events
Keywords: PD-1 inhibitor; Nivolumab; Pembrolizumab; Atezolizumab; Immune-Related Adverse Events; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; Nivolumab; pembrolizumab; atezolizumab; Antineoplastic Agents; Carboplatin; Cisplatin; Vinorelbine; Gemcitabine; Pemetrexed; Docetaxel; Vinblastine; Mitomycin; Gefitinib; Erlotinib Hydrochloride; Afatinib; Crizotinib; ceritinib; alectinib; osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- PD-1 inhibitor: Patients over 18 years of age with a diagnosis of non-small cell lung cancer and being received PD-1 inhibitors as a second line treatment from cytotoxic chemotherapy or as a third line for those received tyrosine kinase inhibitors as a first line, from August 2017 (the first month PD-1 inhibitors were reimbursed in South Korea) to September 2018.
  Interventions: Drug: PD-1 inhibitor
- Chemotherapy Drugs, Cancer: Patients over 18 years of age with a diagnosis of non-small cell lung cancer and being received cytotoxic chemotherapy or tyrosine kinase inhibitors (epidermal growth cell receptor (EGFR) and anaplastic lymphoma kinase (ALK) inhibitors) from August 2017 to September 2018. Each patient switching to PD-1 inhibitor will be matched to three reference standard chemotherapy users.
  Interventions: Drug: Chemotherapy Drugs, Cancer

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 inhibitors are a group of checkpoint inhibitors being developed for the treatment of cancer. PD-1 and PD-L1 are both proteins present on the surface of cells. Immune checkpoint inhibitors such as these are emerging as a front-line treatment for several types of cancer. The investigators will include nivolumab, pembrolizumab, and atezolizumab as PD-1 inhibitors as these drugs are reimbursed by health authority of South Korea.
  Other Names: OPDIVO; KEYTRUDA; TECENTRIQ
  Groups: PD-1 inhibitor
Drug: Chemotherapy Drugs, Cancer — Chemotherapy is a type of pharmacotherapy for cancer, that uses one or more anti-cancer drugs as part of a standardized chemotherapy regimen. The investigators will include cytotoxic chemotherapy and tyrosine kinase inhibitors (epidermal growth cell receptor (EGFR) and anaplastic lymphoma kinase (ALK) inhibitors).
  Other Names: Carboplatin; Cisplatin; Vinorelbine; Gemcitabine; Pemetrexed; Docetaxel; Vinblastine; Mitomycin C; Gefitinib; Erlotinib; Afatinib; Crizotinib; Ceritinib; Alectinib; Osimertinib
  Groups: Chemotherapy Drugs, Cancer

SUMMARY:
The objective of our study is to assess the risk of immune-related adverse events associated with PD-1 inhibitors use compared to standard chemotherapy use in patients with non small cell lung cancer, using nationwide healthcare database.

DETAILED DESCRIPTION:
This observational, retrospective cohort study will evaluate the risk of immune-related adverse events associated with PD-1 inhibitors use compared to standard chemotherapy use in patients with non small cell lung cancer, using nationwide healthcare database. PD-1 inhibitors will be defined as nivolumab, pembrolizumab, and atezolizumab. Standard chemotherapy will be defined as cytotoxic chemotherapy or tyrosine kinase inhibitors (epidermal growth cell receptor (EGFR) and anaplastic lymphoma kinase (ALK) inhibitors). The investigators will assess exposure on the cohort entry using the intention-to-treat approach with the 6-month exposure risk window from the first PD-1 inhibitor prescription to avoid bias from informative censoring. Immune-related adverse events will be defined by using pre-specified algorithms using diagnosis and corticosteroid prescription records (high dose of oral corticosteroids, defined as ≥ 30 mg/day, or systemic corticosteroid injection) to reduce outcome misclassification. The investigators will use a multivariable Cox proportional hazard model to estimate hazard ratio (HR) and 95% confidence intervals (CI). The model will be adjusted for pre-existing autoimmunity, history of lung cancer surgery, radiation therapy, tyrosine kinase inhibitor use, and previous systemic corticosteroid use. All analyses will be undertaken using SAS 9.4 (SAS Institute Inc., Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with lung cancer (ICD-10: C33-C34) between 2017 and 2018.

Exclusion Criteria:

* Individuals less than 18 years of age
* Individuals received any systemic anticancer therapies in 2007
* Having no records of prescription of PD-1 inhibitors or standard chemotherapy at least once between 2017 and 2018
* Individuals received treatments indicated for small cell lung cancer (etoposide, ifosfamide, irinotecan, belotecan, and topotecan) on or before the first date of standard chemotherapy to restrict study subjects to patients with non small cell lung cancer only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be formed by identifying all patients newly treated with standard chemotherapy who subsequently switched to PD-1 inhibitors, from 21 August 2017 to 31 September 2018, with follow-up until 31 December 2018. Patients who remained on standard chemotherapy treatment will be selected as comparators.
Sampling Method: Non-Probability Sample
Enrollment: 4724 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-09-23 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hazard ratio for immune-related adverse events | August 2017 to December 2018
  The ratio of hazard rates of immune-related adverse events in PD-1 inhibitor users vs. standard chemotherapy users

SECONDARY OUTCOMES:
Hazard ratio for eleven subdivided groups of immune-related adverse events by organ class | August 2017 to December 2018
  The ratio of hazard rates of eleven subdivided organ-specific immune-related adverse events (pulmonary, endocrine, cardiovascular, gastrointestinal, hepatic, muscluoskeletal, neurological, ocular, renal, skin, and hematologic) in PD-1 inhibitor users vs. standard chemotherapy users

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Young Shin, PhD, Principal Investigator — Sungkyunkwan University

REFERENCES:
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Postow MA, Sidlow R, Hellmann MD. Immune-Related Adverse Events Associated with Immune Checkpoint Blockade. N Engl J Med. 2018 Jan 11;378(2):158-168. doi: 10.1056/NEJMra1703481. No abstract available. PMID 29320654
- [Background] Baxi S, Yang A, Gennarelli RL, Khan N, Wang Z, Boyce L, Korenstein D. Immune-related adverse events for anti-PD-1 and anti-PD-L1 drugs: systematic review and meta-analysis. BMJ. 2018 Mar 14;360:k793. doi: 10.1136/bmj.k793. PMID 29540345
- [Background] Johnson DB, Sullivan RJ, Menzies AM. Immune checkpoint inhibitors in challenging populations. Cancer. 2017 Jun 1;123(11):1904-1911. doi: 10.1002/cncr.30642. Epub 2017 Feb 27. PMID 28241095
- [Background] Kobayashi K, Nakachi I, Naoki K, Satomi R, Nakamura M, Inoue T, Tateno H, Sakamaki F, Sayama K, Terashima T, Koh H, Abe T, Nishino M, Arai D, Yasuda H, Kawada I, Soejima K, Betsuyaku T; Keio Lung Oncology Group (KLOG). Real-world Efficacy and Safety of Nivolumab for Advanced Non-Small-cell Lung Cancer: A Retrospective Multicenter Analysis. Clin Lung Cancer. 2018 May;19(3):e349-e358. doi: 10.1016/j.cllc.2018.01.001. Epub 2018 Jan 5. PMID 29398578
- [Background] Naidoo J, Wang X, Woo KM, Iyriboz T, Halpenny D, Cunningham J, Chaft JE, Segal NH, Callahan MK, Lesokhin AM, Rosenberg J, Voss MH, Rudin CM, Rizvi H, Hou X, Rodriguez K, Albano M, Gordon RA, Leduc C, Rekhtman N, Harris B, Menzies AM, Guminski AD, Carlino MS, Kong BY, Wolchok JD, Postow MA, Long GV, Hellmann MD. Pneumonitis in Patients Treated With Anti-Programmed Death-1/Programmed Death Ligand 1 Therapy. J Clin Oncol. 2017 Mar;35(7):709-717. doi: 10.1200/JCO.2016.68.2005. Epub 2016 Sep 30. PMID 27646942
- [Background] Remon J, Mezquita L, Corral J, Vilarino N, Reguart N. Immune-related adverse events with immune checkpoint inhibitors in thoracic malignancies: focusing on non-small cell lung cancer patients. J Thorac Dis. 2018 May;10(Suppl 13):S1516-S1533. doi: 10.21037/jtd.2017.12.52. PMID 29951303